CLINICAL TRIAL: NCT00509756
Title: Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of FXR-450 Administered Orally to Healthy Japanese Male Subjects
Brief Title: Study Evaluating FXR-450 in Healthy Japanese Men
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Please see termination statement in the detailed description.
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 3213A1-1002
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2010-10

CONDITIONS: Healthy
Keywords: healthy subjects
MeSH Terms: interventions — WAY-362450

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Drug: FXR-450
  Interventions: Drug: FXR-450
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FXR-450 — capsule, single oral doses from 10 mg to 450 mg
  Arms: 1
Drug: Placebo — capsule similar to active drug
  Arms: 2

SUMMARY:
The primary purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of a single dose of FXR-450 in healthy Japanese men.

DETAILED DESCRIPTION:
This study was terminated on May 2008. The reason for termination was due to pharmacokinetics issues. The decision to terminate was not due to safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 20 to 45 years.
* Healthy as determined by the investigator.
* Nonsmoker or smoker of fewer than 10 cigarettes per day.

Exclusion Criteria:

* A history or active presence of clinically important medical disease.
* Any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the test article (e.g., resection of liver, kidney, gallbladder, or gastrointestinal tract).

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2007-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome is safety and tolerability. | 4 days

SECONDARY OUTCOMES:
Pharmacokinetics | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Tokyo, Tokyo, Japan